CLINICAL TRIAL: NCT05721183
Title: Evaluation of the National Tool for Observation of Infection Prevention Measures in the Healthcare (NOST) - a Cluster Randomized Trial
Brief Title: Evaluation of the National Tool for Observation of Infection Prevention Measures in the Healthcare (NOST)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Norwegian Institute of Public Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NOST
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Infections, Respiratory; Healthcare Worker Patient Transmission
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Intervention Model Description: The intervention is to implement NOST, which includes:
  * observation and recording of compliance with hand hygiene recommendations
  * identification of areas for improvement
  * training or other actions taken to improve IPC in general or compliance with hand hygiene.
  Thus, the intervention includes both observation of compliance and any additional improvement measures initiated as a result of the introduced NOST.
  When the intervention group has implemented and followed NOST for a year, investigators will measure compliance with hand hygiene recommendations and reported HAIs, in wards that have had NOST and in wards that have not introduced NOST.
  The intervention arm will be followed over time with repeated measurements of both compliance with hand hygiene and other outcome measures, to see if the effect increases in line with implemented observations and quality improvement measures, or if the effect decreases during the study period.
Who Masked: Outcomes Assessor
Masking Description: The reserachers who evaluates the outcome of interest will be masked for the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NOST (Experimental): The intervention is to implement NOST, which includes:
  observation and recording of compliance with hand hygiene recommendations identification of areas for improvement training or other actions taken to improve IPC in general or compliance with hand hygiene.
  Thus, the intervention includes both observation of compliance and any additional improvement measures initiated as a result of the introduced NOST.
  When the intervention group has implemented and followed NOST for a year, the investigators will measure compliance with hand hygiene recommendations and reported HAIs, in wards that have had NOST and in wards that have not introduced NOST.
  The intervention arm will be followed over time with repeated measurements of both compliance with hand hygiene and other outcome measures, to see if the effect increases in line with implemented observations and quality improvement measures, or if the effect decreases during the study period.
  Interventions: Behavioral: NOST
- Control (No Intervention): Participants in the no intervention arm arm are asked not to implement NOST.

INTERVENTIONS:
Behavioral: NOST — The intervention is to implement NOST, which includes:
  observation and recording of compliance with hand hygiene recommendations identification of areas for improvement training or other actions taken to improve IPC in general or compliance with hand hygiene.
  Thus, the intervention includes both observation of compliance and any additional improvement measures initiated as a result of the introduced NOST.
  When the intervention group has implemented and followed NOST for a year, the investigators will measure compliance with hand hygiene recommendations and reported HAIs, in wards that have had NOST and in wards that have not introduced NOST.
  The intervention arm will be followed over time with repeated measurements of both compliance with hand hygiene and other outcome measures, to see if the effect increases in line with implemented observations and quality improvement measures, or if the effect decreases during the study period.
  Arms: NOST

SUMMARY:
The Norwegian Institute of Public Health (NIPH) is introducing a new electronic tool for direct observation of compliance with recommended infection prevention and control measures in healthcare. The solution is called the National Tool for Observation of Infection Prevention Measures (NOST). NOST is a quality improvement tool that includes a web-based solution for observing compliance with recommendations for hand hygiene and other IPC measures. Through NOST, healthcare personnel will be able to identify the local level of compliance, which in turn can reveal areas for improvement.

This protocol includes the evaluation of NOST in hospitals. The evaluation is designed as a cluster-randomized controlled trial with two arms where eligible wards in hospitals are randomly allocated into an intervention and a control arm. NOST is implemented in the intervention wards at the start of the evaluation period, and compliance with hand hygiene and other outcomes are measured in both the interventions and control wards one year later.

The objective of evaluating NOST is to:

* measure if implementation of NOST leads to improved infection prevention and control in the form of increased compliance with hand hygiene recommendations, and
* measure if changes in the quality of infection prevention and control as a result of implemented NOST affects the epidemiology of healthcare-associated infections in healthcare institutions and the length of hospital stays.

DETAILED DESCRIPTION:
The evaluation og NOST is designed as a cluster-randomized controlled trial with two arms where eligible wards in hospitals are randomly allocated into an intervention and a control arm. NOST is implemented in the intervention wards at the start of the evaluation period, and compliance with hand hygiene and other outcomes are measured in both the interventions and control wards one year later.

Intervention

The intervention in the study is to implement NOST, which includes:

* observation and recording of compliance with hand hygiene recommendations
* identification of areas for improvement
* training or other actions taken to improve IPC in general or compliance with hand hygiene.

Thus, the intervention includes both observation of compliance and any additional improvement measures initiated as a result of the introduced NOST.

Observations of hand hygiene will be carried out in sessions of 20-30 minutes. During this period, all situations where hand hygiene is indicated (recommended) and whether hand hygiene is performed or not, are recorded. The number of hand hygiene indications during a session varies but will often be between 10 and 20.

When the intervention group has implemented and followed NOST for a year, the investigators will measure compliance with hand hygiene recommendations and reported HAIs, in wards that have had NOST and in wards that have not introduced NOST.

The intervention arm will be followed over time with repeated measurements of both compliance with hand hygiene and other outcome measures, to see if the effect increases in line with implemented observations and quality improvement measures, or if the effect decreases during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Hospital wards with day- and night care.

Exclusion Criteria:

* Intensivecare units.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2023-02-20 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Hand hygiene observations | Day 1 to one year later
  Self-reported proportion of correct compliance, in total and by occupation

SECONDARY OUTCOMES:
Outbreaks of infectious diseases | Day 1 to one year later
  Proportion of outbreaks per ward and secondary attack rate by inpatients and staff. Data collected from VESUV
Surveillance of healthcare-associated infections | Day 1 to one year later
  Proportion of infected inpatients by type of infections. Data collected from NOIS
Surveillance of postoperative site infections | Day 1 to one year later
  Proportion of infected patients by type of surgery and type of infections. Data collected from NOIS and POSI
Length of stay | Day 1 to one year later
  Mean and median bed-days per stay. Data collected from NRP

CONTACTS AND LOCATIONS:
Overall Officials: Petter Elstrøm, PhD, Principal Investigator — Norwegian Institute of Public Health
Locations (1):
- Norwegian Institute of Public Health, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
In this project, the investigators will not register or collect direct identifiable personal data. In the hand hygiene observations, only the events and occupation are recorded, but not personal data on the people observed. Furthermore, the investigators will only ask for statistics from VESUV and NOIS/NOIS-POSI. This data will include the number of people infected in outbreaks per ward distributed by employees and inpatients, as well as the number of inpatients with relevant types of infection in the surveillance of HAI. These data are regularly published at the hospital level. The investigators will apply for data from NPR that includes information on each patient admitted to the relevant wards in the period from 1 January 2022 to mid-2024. However, the investigators will ask for data without directly personally identifiable information (data without name and social security number).